CLINICAL TRIAL: NCT04092621
Title: Rapid Atrial Fibrillation Treatment Strategy
Acronym: RAFTS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Our Lady of the Lake Hospital (Other)
Responsible Party: Principal Investigator, Hollis O Neal, Medical Director of Research, Our Lady of the Lake Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-106
Record Dates: First submitted 2019-09-06; First posted 2019-09-17 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: New Onset Atrial Fibrillation; Sepsis; Respiratory Failure
Keywords: new onsent atrial fibrillation; sepsis; critical care; direct current cardioversion; atrial fibrillation treatment
MeSH Terms: conditions — Sepsis; Respiratory Insufficiency | interventions — Amiodarone; Injections; Electric Countershock

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Rhythm-control strategy (Experimental): The patient will receive 1) amiodarone 150mg bolus over ten minutes followed by intravenous (IV) 1mg/min for 6 hours and then 0.5mg/min for 18hours, and 2) direct current cardioversion (DCC) at the completion of initial 6 hour IV bolus or within 24 hours of new onset of atrial fibrillation. Patient will be placed on by mouth amiodarone 400mg three times daily for seven days, then 400mg twice daily for seven days, then 400mg once daily for seven days, then 200mg daily until stop date which will be by provider discretion after discharge from ICU. If the patient does not convert to a normal sinus rhythm with routine DCC then they will remain in the rhythm-control strategy to receive amiodarone as directed. Amiodarone may be extended at discretion of provider for 30 days with discontinuation if adverse effects. If no contraindications, anticoagulation will be recommended prior to DCC with enoxaparin 1mg/kg every 12 hours.
  Interventions: Drug: Amiodarone in Parenteral Dosage Form; Drug: Amiodarone Pill; Procedure: Direct Current Cardioversion (DCC)
- Rate-control strategy (Active Comparator): At treating physician's discretion, one of the following, or a combination of the following, will be administered to the patient: Amiodarone, beta blockers or non-dihydropyridine calcium channel blockers, digoxin. The target heart rate is less than 120 beats per minute (bpm) or maintained hemodynamics. Patients in the rate-control arm who are hypotensive after new onset atrial fibrillation can undergo DCC at the provider's discretion and crossover into the rhythm-control arm.
  Interventions: Drug: Rate-control therapy

INTERVENTIONS:
Drug: Amiodarone in Parenteral Dosage Form — Amiodarone IV
  Other Names: Cordarone
  Arms: Rhythm-control strategy
Drug: Amiodarone Pill — Amiodarone tablet
  Other Names: Cordarone
  Arms: Rhythm-control strategy
Procedure: Direct Current Cardioversion (DCC) — Convert arrhythmia back to sinus rhythm
  Arms: Rhythm-control strategy
Drug: Rate-control therapy — one or combination of the following: Amiodarone, beta blockers or non-dihydropyridine calcium channel blockers, digoxin
  Arms: Rate-control strategy

SUMMARY:
Prospective, randomized, open-label clinical trial studying the treatment of new onset atrial fibrillation in critically ill patients with septic shock. Patients will be assigned to rhythm vs rate control strategies with various outcome measures assessed.

DETAILED DESCRIPTION:
Data have demonstrated that critically ill patients with septic shock who develop atrial fibrillation suffer a greater likelihood of death and other complications when compared with patients who remain in sinus rhythm, however, little evidence exists to inform treatment strategies in this population. Ours is a pilot study evaluating rhythm vs rate control strategies in patients with septic shock and respiratory failure requiring invasive mechanical ventilation who develop new onset atrial fibrillation (NOAF). Design will be prospective, randomized, open-label. Patients in the rhythm control arm will receive IV amiodarone infusion followed by attempt at electrical cardioversion within 24 hours development of NOAF. Those in the rate control arm will receive negative chronotropic agents (beta blockers, calcium channel blockers, amiodarone, or digoxin) at the discretion of the treating physician. Available patient data will be collected for a total of 180 days following enrollment, and outcomes assessed will include ICU length of stay, ventilator free days, and time on vasopressors

ELIGIBILITY:
Inclusion Criteria:

* No history of atrial fibrillation
* Meet Sepsis-3 criteria
* New onset atrial fibrillation in the ICU
* Atrial fibrillation treatment warranted
* Anticoagulation therapy not contraindicated
* On a ventilator
* Patient or family member willing to provide informed consent to participate in study

Exclusion Criteria:

* Post-cardiac or thoracic surgery
* Hemodynamically unstable
* Unable to tolerate anticoagulation
* Physician provider does not agree for patient to participate in study
* Patient or family member unwilling or unable to provide informed consent
* Expected death within 24 hours
* Non-English speakers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-09-16 (Estimated); Primary Completion 2020-09-15 (Estimated); Study Completion 2020-09-15 (Estimated)

PRIMARY OUTCOMES:
ICU Length of Stay (LOS) | 28 days
  Number of days patient was in the ICU
Ventilation-free days | 28 days
  Days alive and free from mechanical ventilation
Vasopressor days | 28 days
  If vasopressors are administered, number of days patient received vasopressors in the ICU

CONTACTS AND LOCATIONS:
Overall Officials: Hollis R O'Neal, MD, Principal Investigator — Louisiana State University Health Sciences Center
Locations (1):
- Our Lady of the Lake Regional Medical Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Meierhenrich R, Steinhilber E, Eggermann C, Weiss M, Voglic S, Bogelein D, Gauss A, Georgieff M, Stahl W. Incidence and prognostic impact of new-onset atrial fibrillation in patients with septic shock: a prospective observational study. Crit Care. 2010;14(3):R108. doi: 10.1186/cc9057. Epub 2010 Jun 10. PMID 20537138
- [Background] Yoshida T, Fujii T, Uchino S, Takinami M. Epidemiology, prevention, and treatment of new-onset atrial fibrillation in critically ill: a systematic review. J Intensive Care. 2015 Apr 23;3(1):19. doi: 10.1186/s40560-015-0085-4. eCollection 2015. PMID 25914828
- [Background] Caldeira D, David C, Sampaio C. Rate versus rhythm control in atrial fibrillation and clinical outcomes: updated systematic review and meta-analysis of randomized controlled trials. Arch Cardiovasc Dis. 2012 Apr;105(4):226-38. doi: 10.1016/j.acvd.2011.11.005. Epub 2012 Jan 21. PMID 22633297
- [Background] Chean CS, McAuley D, Gordon A, Welters ID. Current practice in the management of new-onset atrial fibrillation in critically ill patients: a UK-wide survey. PeerJ. 2017 Sep 8;5:e3716. doi: 10.7717/peerj.3716. eCollection 2017. PMID 28929012
- [Background] Sibley S, Muscedere J. New-onset atrial fibrillation in critically ill patients. Can Respir J. 2015 May-Jun;22(3):179-82. doi: 10.1155/2015/394961. PMID 26057373
- [Background] Walkey AJ, Hogarth DK, Lip GYH. Optimizing atrial fibrillation management: from ICU and beyond. Chest. 2015 Oct;148(4):859-864. doi: 10.1378/chest.15-0358. PMID 25951122
- [Background] Kanji S, Williamson DR, Yaghchi BM, Albert M, McIntyre L; Canadian Critical Care Trials Group. Epidemiology and management of atrial fibrillation in medical and noncardiac surgical adult intensive care unit patients. J Crit Care. 2012 Jun;27(3):326.e1-8. doi: 10.1016/j.jcrc.2011.10.011. Epub 2012 Jan 4. PMID 22226423
- [Background] Mayr A, Ritsch N, Knotzer H, Dunser M, Schobersberger W, Ulmer H, Mutz N, Hasibeder W. Effectiveness of direct-current cardioversion for treatment of supraventricular tachyarrhythmias, in particular atrial fibrillation, in surgical intensive care patients. Crit Care Med. 2003 Feb;31(2):401-5. doi: 10.1097/01.CCM.0000048627.39686.79. PMID 12576943
- [Background] Walkey AJ, Greiner MA, Heckbert SR, Jensen PN, Piccini JP, Sinner MF, Curtis LH, Benjamin EJ. Atrial fibrillation among Medicare beneficiaries hospitalized with sepsis: incidence and risk factors. Am Heart J. 2013 Jun;165(6):949-955.e3. doi: 10.1016/j.ahj.2013.03.020. Epub 2013 Apr 25. PMID 23708166
- [Background] Arrigo M, Jaeger N, Seifert B, Spahn DR, Bettex D, Rudiger A. Disappointing Success of Electrical Cardioversion for New-Onset Atrial Fibrillation in Cardiosurgical ICU Patients. Crit Care Med. 2015 Nov;43(11):2354-9. doi: 10.1097/CCM.0000000000001257. PMID 26468695
- [Background] Walkey AJ, Wiener RS, Ghobrial JM, Curtis LH, Benjamin EJ. Incident stroke and mortality associated with new-onset atrial fibrillation in patients hospitalized with severe sepsis. JAMA. 2011 Nov 23;306(20):2248-54. doi: 10.1001/jama.2011.1615. Epub 2011 Nov 13. PMID 22081378
- [Result] Liu WC, Lin WY, Lin CS, Huang HB, Lin TC, Cheng SM, Yang SP, Lin JC, Lin WS. Prognostic impact of restored sinus rhythm in patients with sepsis and new-onset atrial fibrillation. Crit Care. 2016 Nov 18;20(1):373. doi: 10.1186/s13054-016-1548-2. PMID 27855722